CLINICAL TRIAL: NCT06137755
Title: A Multicenter, Active-controlled, Open-label Phase I Study to Assess Safety and Tolerability and to Explore Immunogenicity of CVI-VZV-001 Vaccine in Healthy Adults Aged 50 to 64 Years
Brief Title: Safety and Immunogenicity of CVI-VZV-001 for Prevention of Herpes Zoster in Healthy Adults Age 50 Years and Above
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CHA Vaccine Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CVI-VZV-001-CT2101
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Vaccine-Preventable Diseases; Herpes Zoster
MeSH Terms: conditions — Vaccine-Preventable Diseases; Herpes Zoster

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Recombinant Herpes Zoster Vaccine(CVI-VZV-001) 0.37 mL per dose, Intramuscular injection at Baseline, Week 8 / total 2 doses
  Interventions: Biological: CVI-VZV-001
- Group 2 (Experimental): Recombinant Herpes Zoster Vaccine(CVI-VZV-001) 0.50 mL per dose, Intramuscular injection at Baseline, Week 8 / total 2 doses
  Interventions: Biological: CVI-VZV-001
- Group 3 (Experimental): Recombinant Herpes Zoster Vaccine(CVI-VZV-001) 0.75 mL per dose, Intramuscular injection at Baseline, Week 8 / total 2 doses
  Interventions: Biological: CVI-VZV-001
- Active Control (Active Comparator): Shingrix 0.50 mL per dose, Intramuscular injection at Baseline, Week 8 / total 2 doses
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: CVI-VZV-001 — Investigational Product
  Arms: Group 1; Group 2; Group 3
Biological: Shingrix — Investigational Product
  Arms: Active Control

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the investigational medicinal product, CVI-VZV-001.

DETAILED DESCRIPTION:
A Multicenter, Active-controlled, Open-label Phase I Study to Assess Safety and Tolerability and to Explore Immunogenicity of CVI-VZV-001 Vaccine in Healthy Adults Aged 50 to 64 Years

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over 50 years old and under 65 years old
2. Those who voluntarily decided to participate and gave written consent after hearing and understanding the detailed explanation of this clinical trial
3. Women with childbearing potential and those who agree to use the contraceptive method* permitted up to 3 months after the final vaccination for clinical trials (* Combination use such as hormonal contraception, intrathyroidal device (IUD (Intrauterine device) or IUS (Intrauterine system), vasectomy, tubal stomy, double block method (cervical cap, use with contraceptive diaphragm)
4. Women of childbearing potential with negative result at pregnancy test before vaccination for clinical trials.

Exclusion Criteria:

1. Those with a past history of shingles before screening
2. Persons with hypersensitivity to clinical investigational products or the ingredients of clinical investigational products
3. Those with thrombocytopenia or other coagulation disorders who should not receive intramuscular injections, or those receiving anticoagulant therapy*

   *Anticoagulant therapy: Continuous use of anticoagulants such as coumarin/warfarin or new oral anticoagulants/antiplatelet agents
4. Those with a history of immune dysfunction, including immunodeficiency disease
5. Those suffering from chronic underlying diseases that, in the opinion of the investigator, may interfere with the progress and completion of this clinical trial
6. Those with a history of excessive alcohol consumption or drug addiction
7. Persons with a history of serious adverse events, allergies or hypersensitivity reactions related to vaccination (e.g. anaphylaxis, Guillain-Barré Syndrome)
8. Those with a history of malignant tumor
9. Those who developed a fever (tympanic membrane temperature of 38.0°C or higher) within 3 days prior to the first vaccination of clinical investigational product, suffered from a febrile illness on the day of vaccination, or suffered from a disease with moderate or more acute symptoms (mild illness without fever) (e.g. If you have mild diarrhoea, mild upper respiratory infection), you can participate in the clinical trial at the discretion of the investigator.)
10. Those who have received chickenpox or shingles vaccine before screening
11. Those who have participated in past chickenpox or shingles vaccine clinical trials
12. Those who have been vaccinated with another vaccine within 4 weeks prior to the first injection of the investigational product, or who plan to be vaccinated with another vaccine by 48 weeks after the second injection of the investigational product (however, seasonal or pandemic flu) (inactivated and subunit influenza vaccine and COVID-19 vaccine for prevention of flu) are contraindicated only within 2 weeks before and after vaccination of each clinical investigational product)
13. Those who have received blood products or immunoglobulin within 3 months prior to receiving the first clinical investigational product, or those who plan to administer it during the clinical trial period
14. Those who have received immunosuppressants, immunomodulating drugs, other cytotoxic anticancer drugs that may affect immunity, or have experienced radiation therapy within 6 months prior to receiving the first clinical investigational product.
15. Those who have experienced systemic steroid administration within 3 months prior to receiving the first clinical investigation drug (those who are taking a dose of 20 mg/day or more based on prednisone continuously for more than 2 weeks) However, topical, inhalation ( Inhaled, intranasal, intra-articular, and intra-bursal administration is permitted regardless of dosage.
16. Organ transplant or hematopoietic stem cell transplant patients
17. Those with positive virus test results (HCV Ab, HBsAg, HIV Ab) performed at screening
18. Persons with clinically significant abnormalities in tests performed during screening (clinical laboratory tests, electrocardiogram, vital signs, etc.)
19. Those taking antiviral drugs (Acyclovir, Valacyclovir, Famciclovir, Ganciclovir, etc.) known to be effective against varicella-zoster virus at the time of screening (topical use of antiviral drugs is permitted)
20. Those with a history of active tuberculosis
21. A person who has received another clinical investigational product or applied a clinical trial medical device within 6 months before participating in a clinical trial
22. Pregnant or lactating women
23. If the investigator determines that the subject is unsuitable for this clinical trial for other reasons

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Immediate adverse events | within 30 minutes at each vaccination timepoint
  Occurrence of immediate adverse events
Solicited local and systemic signs and symptoms | Day 0 - Day 6 for each vaccination timepoint
  Occurrence, severity, and duration of solicited local injection site reactions for 7 days (Day 0-Day 6) following each vaccination. (i.e., pain, redness, swelling)
  Occurrence, severity, and duration of solicited systemic reactions for 7 days (Day 0-Day 6) following each vaccination. (i.e., myalgia, fatigue, headache, chills, fever)
Unsolicited signs and symptoms | Until Week 4 post the 2nd vaccination
  Occurrence, severity, and relationship to vaccination of unsolicited adverse events until 28 days following the last vaccination
SAEs | Until Week 48 post the 2nd vaccination
  Occurrence of serious adverse events (SAEs)
MAAEs | Until Week 48 post the 2nd vaccination
  Occurrence of Medically attended adverse events(MAAEs)
AESIs | Until Week 48 post the 2nd vaccination
  Occurrence of adverse events (AEs) of special interest
Safety as measured by clinical laboratory test, vial sign and physical examination parameters | Until Week 4 post the 2nd vaccination
  Occurrence, intensity, and relationship to vaccination of clinically significant adverse events

SECONDARY OUTCOMES:
Humoral immune response before the first and second vaccinations of investigational drugs and at 4, 24, and 48 weeks after the second vaccination. | Pre vaccinations(Day0, week 8) of 1st and 2nd vaccination, and at 4, 24, and 48 weeks post the 2nd vaccination
  Anti-VZV antibody titer, Anti-VZV glycoprotein ELISA
Cell-mediated immunity (CMI) immune response before the first and second vaccinations of investigational drugs and at 4, 24, and 48 weeks after the second vaccination. | Pre vaccinations(Day0, week 8) of 1st and 2nd vaccination, and at 4, 24, and 48 weeks post the 2nd vaccination
  IFN-gamma ELISpot, Polyfunctional T cell(ICS)

CONTACTS AND LOCATIONS:
Overall Officials: Jeonghyeon Choi, Principal Investigator — The Catholic University of Korea Eunpyeong St. Mary's Hospital
Locations (2):
- South Korea (2):
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu
  - Bundang CHA General Hospital, Seongnam-si, Gyeonggi-do